CLINICAL TRIAL: NCT03201133
Title: Clinical Subgroups Identification in Patellofemoral Pain Syndrome Patients
Brief Title: Clinical Subgroups in Patellofemoral Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Other Study IDs: UFRGS 1.978.838
Record Dates: First submitted 2017-06-21; First posted 2017-06-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patellofemoral pain syndrome with changes in proximal factors
  Interventions: Diagnostic Test: Neuromuscular evaluation
- Patellofemoral pain syndrome with changes in local factors
  Interventions: Diagnostic Test: Neuromuscular evaluation
- Patellofemoral pain syndrome with changes in distal factors
  Interventions: Diagnostic Test: Neuromuscular evaluation

INTERVENTIONS:
Diagnostic Test: Neuromuscular evaluation — (1) Muscle trunk endurance test; (2) Hip isometric strength (abductor, lateral rotation, extension); (3) Knee extensor isometric strength; (4) unilateral squat; (5) navicular drop test; (6) muscle architecture at rest of gluteus medius, gluteus maximus,vastus lateralis, vastus medialis and rectus femoris; (7) muscle activation during unilateral squat (gluteus and quadriceps muscles); (8) pennation angle of obliques vastus medialis; (9) medial patellofemoral ligament length; (10) knee pain.

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a multifactorial pathology characterized by diffuse retropatellar and peripatellar pain in the knee joint, exacerbated by overloading activities on the patellofemoral joint. However, this disease showed high degree of patients not responsive to therapeutic strategies. This condition occurred because several factors is related to disease such as: (1) proximal factors (involving trunk and hip), (2) local factors (surrounding and or within the patellofemoral joint) and (3) distal factors (involving ankle and foot). Thus, the identification of clinical subgroups based in anatomic changes (proximal, local and distal factors) is a recent strategy that could help in the therapeutic strategies focused on the etiology of the disease, improve responsiveness to treatment, clinical and functional benefits.

ELIGIBILITY:
Inclusion Criteria:

* Peripatellar or retropatellar pain in at least two of the following situations: squatting, running, kneeling, jumping, climbing or descending stairs and sitting for a prolonged period of time for at least three months.

Exclusion Criteria:

* Engaged in systematic exercise with focus on lower limb in the last six months and Had an injury to the hip and ankle joint in the last 12 months.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patellofemoral pain syndrome women
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Muscular strength tests of hip and knee muscles. | 1 day
  Isometric torque of knee extensor muscles, hip abductor, extension and medial rotation muscles through hand-held dynamometer tests will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.
Muscle thickness measures | 1 day
  Muscle thickness (in millimeters) of vastus lateralis, vastus medialis and rectus femoris muscle. Muscle thickness of gluteus medius, maximus and peroneus muscle through ultrasound equipment. Tests Test will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.
Muscle activation of knee, hip and foot muscles | 1 day
  Muscle activation measures of quadriceps, gluteus maximus, gluteus medius and peroneus muscles during unilateral squat through surface electromyography. Tests will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.
Kinematics during unilateral squat | 1 day
  Pelvis, hip, knee and ankle angular displacement during unilateral squat through kinematics analysis. Tests will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.
Fascicle length measures | 1 day
  Fascicle length (in milimeters) of vastus lateralis, vastus medialis and rectus femoris muscle through ultrasound equipment. Tests Test will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.
Pennation angle measures | 1 day
  Pennation angle (in °) of vastus lateralis, vastus medialis and rectus femoris muscle through ultrasound equipment. Tests Test will be performed to create clinical subgroups after cluster analysis for a focused intervention in the second step.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Research Laboratory, Pôrto Alegre, Rio Grande do Sul, Brazil